CLINICAL TRIAL: NCT00073190
Title: Randomized Controlled Testing of Osteoporosis Education
Brief Title: Patient- and Physician-Based Osteoporosis Education
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Arthritis Foundation (Other)
Responsible Party: Principal Investigator, Daniel H. Solomon, M.D.,MPH, Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: K23AR048616 (NIH); K23AR048616 (NIH); NIAMS-074
Record Dates: First submitted 2003-11-17; First posted 2003-11-18 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Osteoporosis; Osteoporosis, Postmenopausal
Keywords: Patient Education; Physician Education
MeSH Terms: conditions — Osteoporosis; Osteoporosis, Postmenopausal

INTERVENTIONS:
Behavioral: Osteoporosis Education

SUMMARY:
Osteoporosis is an important public health problem. Osteoporosis can cause serious health complications and death and leads to increased medical costs. The purpose of this study is to identify an effective method of educating patients and health care professionals about the diagnosis and treatment of osteoporosis.

DETAILED DESCRIPTION:
Osteoporosis affects a large and growing proportion of the population. Multiple drugs for the prevention and treatment of osteoporosis have been developed, tested, and proven effective in the last decade. However, these drugs may not always be adequately prescribed. Several effective nonpharmacological measures also exist for preventing fractures; strength and gait training, home safety modifications, and other lifestyle modifications have all been shown in carefully conducted trails to reduce the risk of falls that lead to osteoporotic fractures. Yet these interventions are under-utilized. Practical public health strategies are needed to bring these experimental findings to widespread use in typical populations of at-risk patients. This study will evaluate innovative fracture prevention interventions targeted to both patients and doctors. Specifically, the study will compare the effects of the patient and physician behavior change intervention alone and in combination on prescribing patterns for osteoporosis therapies and will examine the interventions' effects on fracture prevention behaviors other than medication use.

The patient intervention will consist of two mailings and will be targeted using clinical and demographic data from the State of Pennsylvania's Pharmaceutical Assistance Contract for the Elderly (PACE) and Medicare databases. The first mailing will introduce the topic of osteoporosis and explain why osteoporosis is an important topic for all those receiving the mailing. The second mailing, sent the following month, will reinforce the first mailing and contain patient-specific information based on demographic and clinical factors. This mailing will also focus on several proven prevention strategies, including strength and gait training, vision care, home safety improvements, calcium intake, and pharmaceutical enhancement of bone density.

The physician intervention will be multifaceted and will include a mailed practice audit and one-on-one education through academic detailing. The mail audit will contain information on the physician's PACE patients and an assessment of their osteoporosis risk based on clinical and drug data. Following the mailing, an academic detailer will meet with the physicians receiving the intervention.

Outcome measures will include questionnaires, medication use, Dual Energy X-ray Absorptiometry (DEXA) scans, and use of physical therapy.

ELIGIBILITY:
Inclusion Criteria For Patients:

* PACE beneficiaries who filled at least one prescription for a drug of any type in the year prior to the study
* At high risk for osteoporosis: women and men 75 years or older, patients taking glucocorticoids or psychoactive medications, patients diagnosed with rheumatoid arthritis, and patients with a past fracture
* Have had an outpatient visit with a participating doctor based on Medicare outpatient claims

Inclusion Criteria For Physicians:

* Primary prescribing physicians for PACE beneficiaries

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30000
Dates: Start 2003-09; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H. Solomon, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Daniel H. Solomon MD, MPH, Boston, Massachusetts, United States

REFERENCES:
- [Background] Solomon DH, Finkelstein JS, Katz JN, Mogun H, Avorn J. Underuse of osteoporosis medications in elderly patients with fractures. Am J Med. 2003 Oct 1;115(5):398-400. doi: 10.1016/s0002-9343(03)00357-7. No abstract available. PMID 14553876
- [Background] Solomon DH, Katz JN, La Tourette AM, Coblyn JS. Multifaceted intervention to improve rheumatologists' management of glucocorticoid-induced osteoporosis: a randomized controlled trial. Arthritis Rheum. 2004 Jun 15;51(3):383-7. doi: 10.1002/art.20403. PMID 15188323
- [Background] Warsi A, Wang PS, LaValley MP, Avorn J, Solomon DH. Self-management education programs in chronic disease: a systematic review and methodological critique of the literature. Arch Intern Med. 2004 Aug 9-23;164(15):1641-9. doi: 10.1001/archinte.164.15.1641. PMID 15302634